CLINICAL TRIAL: NCT03794024
Title: Single Center, Randomized Prospective Comparative Effectiveness Study of Dorsal Column Spinal Cord Stimulation to Dorsal Root Ganglion Stimulation in the Treatment of Complex Regional Pain Syndrome
Brief Title: Comparison of Dorsal Column Stimulation to Dorsal Root Ganglion Stimulation for Complex Regional Pain Syndrome
Status: Terminated | Type: Observational
Why Stopped: Manufacturer of the device filed for bankruptcy
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 18-1115
Record Dates: First submitted 2018-12-31; First posted 2019-01-04 (Actual); Results first posted 2020-06-24 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Complex Regional Pain Syndrome
MeSH Terms: conditions — Complex Regional Pain Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Dorsal Column Stimulation: Subjects with Complex Regional Pain Syndrome receiving implant with the Nuvectra Algovita Dorsal Column Spinal Cord Stimulator
  Interventions: Device: The Nuvectra Algovita Dorsal Column Spinal Cord Stimulator
- Dorsal Root Ganglion Stimulation: Subjects with Complex Regional Pain Syndrome receiving implant with the Axium Neurostimulator System
  Interventions: Device: The Axium Neurostimulator System

INTERVENTIONS:
Device: The Nuvectra Algovita Dorsal Column Spinal Cord Stimulator — The Nuvectra Algovita Dorsal Column Spinal Cord Stimulator is indicated as an aid in the management of chronic intractable pain of the trunk and/or limbs, including unilateral or bilateral pain associated with failed back surgery syndrome, intractable low back pain and leg pain.
  Groups: Dorsal Column Stimulation
Device: The Axium Neurostimulator System — The Axium Neurostimulator System is indicated for spinal column stimulation via epidural and intra-spinal lead access to the dorsal root ganglion as an aid in the management of moderate to severe chronic intractable pain of the lower limbs in adult patients with Complex Regional Pain Syndrome Types I and II
  Groups: Dorsal Root Ganglion Stimulation

SUMMARY:
Complex Regional Pain Syndrome (CRPS) is a constellation of pain symptoms which are associated with impairment in mood, social and physical function. Spinal Cord Stimulation (SCS), a technique of placing electrodes into the epidural space is a validated treatment for Complex Regional Pain Syndrome . Treatment of CRPS with SCS, in combination with physical therapy, reduced pain to a greater degree than physical therapy alone. 40%-50% of CRPS patients achieve >50% pain relief with SCS using dorsal column stimulation . Dorsal Root Ganglion (DRG) SCS has also recently demonstrated clinical efficacy in patients with CRPS and peripheral causalgia . The hypothesis is that DRG stimulation is non-inferior to dorsal column SCS in patients with CRPS who have failed to respond to a course of analgesics and physical therapy. The aim to assess functional, quality of life, patient satisfaction and medication requirements in subjects treated with neuromodulation for CRPS and contrast outcomes amongst subjects treated with DRG SCS and dorsal column SCS.

DETAILED DESCRIPTION:
The purpose of this study is to compare outcomes between dorsal column spinal cord stimulation and dorsal root ganglion spinal cord stimulation in patients with Complex Regional Pain Syndrome at an infraumbilical location who have failed a course of conservative management including analgesic pharmacotherapy and physical therapy.

This is a prospective randomized post-marketing clinical study. Patients will be randomized in a 1:1 ratio to Dorsal Column or Dorsal Root Ganglion Spinal Cord Stimulation if they have failed a course of conservative management including analgesics and physical therapy. All patients are expected to undergo clinical, neurological, and imaging assessments, if appropriate, at selected follow-up visits.

The study will be conducted a single center with a target maximum of 62 patients (31 randomized to each group).

Enrollment of subjects in this study is anticipated to take 24 months. Clinical follow-up evaluations will be conducted at 10 days, 1, 3 and 6 months post-implant. The total study duration is expected to be at least 30 months.

All patients presenting to the Investigators with Budapest criteria, research subset , for the diagnosis of Complex Regional Pain Syndrome at an infraumbilical location who have not had an adequate response to a course of conservative management including analgesics and physical therapy will be screened for eligibility. A Screening/Enrollment Log will be utilized in order to maintain a cumulative tracking of all screened patients.

Patients must meet all inclusion/exclusion criteria for enrollment in the clinical study. Reasons for screening failure(s) will be documented.

ELIGIBILITY:
Inclusion Criteria:

* • Patient is greater than18 years of age

  * An infraumbilical location of the index pain
  * Symptoms have been present for greater than 6 months
  * Continuing pain which is disproportionate to any inciting event
  * Report hyperesthesia and/or allodynia
  * Report vasomotor changes including temperature asymmetry and/or skin color changes and/or skin color asymmetry
  * Report edema and/or sweating changes and/or sweating asymmetry
  * Report decreased range of motion and/or motor dysfunction (weakness, tremor, dystonia) and/or trophic changes (hair, nail, skin)
  * Display at least one sign in two or more of the following categories:

    * Sensory: Evidence of hyperalgesia (to pinprick) and/or allodynia (to light touch and/or temperature sensation and/or deep somatic pressure and/or joint movement)
    * Vasomotor: Evidence of temperature asymmetry (>1°C) and/or skin color changes and/or asymmetry
    * Sudomotor/Edema: Evidence of edema and/or sweating changes and/or sweating asymmetry
    * Motor/Trophic: Evidence of decreased range of motion and/or motor dysfunction (weakness, tremor, dystonia) and/or trophic changes (hair, nail, skin)
  * Patient failed to have resolution of symptoms despite at least 4 weeks of conservative management including analgesic pharmacotherapy and physical therapy
  * Patient has index site pain > spine pain
  * The subject is physically and mentally able to participate in the study
  * Patient is willing and able to provide informed consent
  * Patient is willing and able to comply with the study protocol

Exclusion Criteria:

* Previous surgery to the spine which could compromise placement of the study device
* Anatomical spinal abnormality including severe central canal stenosis or bony foraminal impingement which could preclude device placement
* Foreseen need for MRI to monitor or evaluate another chronic condition
* Previous experience with an implanted or trial neuromodulation system (spinal cord stimulation, peripheral nerve stimulation) for the treatment of pain at the index location
* Active local or systemic infection
* Actively in litigation for pain symptoms
* Currently on Workman's Compensation
* Women who are pregnant or intend to become pregnant during the study duration

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with Budapest criteria (research diagnostic definition) of Complex Regional Pain Syndrome occurring below the umbilicus who have not had an adequate response to conservative management including analgesic and physical therapies.
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2020-03-03 (Actual); Study Completion 2020-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bolash, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Roberta Johnson, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dorsal Column Stimulation | Dorsal Root Ganglion Stimulation
Started | 1 | 0
Completed | 0 | 0
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Population: No patients enrolled were randomized into the Dorsal Root Ganglion Stimulation arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dorsal Column Stimulation | Dorsal Root Ganglion Stimulation | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 1 |  | 1
  >=65 years | 0 |  | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 |  | 1
  Male | 0 |  | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  | 0
  Not Hispanic or Latino | 1 |  | 1
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Numerical Rating Scale for Pain Intensity
Description: To compare the outcomes of dorsal column stimulation with Dorsal Root Ganglion stimulation in patients with Complex Regional Pain Syndrome that persist despite a course of conservative management including physical therapy and analgesic pharmacotherapy using an 11-point [0-10] Numerical Rating Scale (NRS) for Pain Intensity at 6 months. A score of zero indicates no pain, and 10 indicates the worst possible pain imaginable.
Time Frame: 6 Months
Population: No patients achieved the 6 month endpoint
Arm/Group | Dorsal Column Stimulation | Dorsal Root Ganglion Stimulation
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change in Oswestry Disability Index for Pain Intensity
Description: To compare the outcomes of dorsal column stimulation with Dorsal Root Ganglion stimulation in patients with Complex Regional Pain Syndrome that persist despite a course of conservative management including physical therapy and analgesic pharmacotherapy in function based on Oswestry Disability Index (ODI) for functional impairment. A score of 0 on the 101-point [0-100] Oswestry Disability Index indicates no disability while 100 indicates bed-bound.
Time Frame: 6 Month
Population: Data were not collected
Arm/Group | Dorsal Column Stimulation | Dorsal Root Ganglion Stimulation
Number analyzed (Participants) | 0 | 0

3. Other Pre Specified Outcome: Change in European Quality of Life 5 Dimension Scale
Description: Change in Quality of Life as measured by the European Quality of Life 5 Dimension (EQ-5D) Scale. The EQ-5D-5L is composed of - the EQ-5D-5L descriptive system and the EQ Visual Analogue scale (EQ VAS). The descriptive system comprises 5 dimensions (mobility, self care, usual activities, pain/discomfort, anxiety/depression). Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. Each level corresponds to 1-digit number expressing the level selected for that dimension.
Time Frame: 6 Months
Population: Data were not collected
Arm/Group | Dorsal Column Stimulation | Dorsal Root Ganglion Stimulation
Number analyzed (Participants) | 0 | 0

4. Other Pre Specified Outcome: Health Status Measured by Short Form-36 (SF-36)
Description: Change in Health Status measured by Short Form-36 (SF-36). This form measures patient's overall health. Scores range from 0 - 100 with lower scores indicating more disability while higher scores indicate less disability.
Time Frame: 6 Months
Population: Data were not collected
Arm/Group | Dorsal Column Stimulation | Dorsal Root Ganglion Stimulation
Number analyzed (Participants) | 0 | 0

5. Other Pre Specified Outcome: Pain Medication Usage
Description: The opioid morphine equivalent conversion factor is used to standardized opioid usage having as a reference morphine as the main indicator for analgesic potency. Oral morphine equivalents are based on the idea that different doses of different opioids may give a similar analgesic effect. Where the doses of two different opioids are considered to give a comparable analgesic effect, they are deemed to be equianalgesic doses.
Time Frame: 6 Months
Population: Data were not collected
Arm/Group | Dorsal Column Stimulation | Dorsal Root Ganglion Stimulation
Number analyzed (Participants) | 0 | 0

6. Other Pre Specified Outcome: Satisfaction With the Pain Relief
Description: There will be 3 separate questions on the form. Subjects will be asked to rate their satisfaction with the pain relief, satisfaction with the therapy in general and their likelihood undergoing the therapy again for a similar outcome as a percentage from 0-100% with 0% indicating no satisfaction/likelihood and 100% indicating completely satisfied and 100% likelihood of undergoing the therapy again for a similar outcome.
Time Frame: 6 Months
Population: Data were not collected
Arm/Group | Dorsal Column Stimulation | Dorsal Root Ganglion Stimulation
Number analyzed (Participants) | 0 | 0

7. Other Pre Specified Outcome: Adverse Events Related to the Procedure or Devices
Description: Descriptive safety data defined as adverse events related to the procedure or devices will be enumerated.
Time Frame: 6 Months
Population: Data were not collected
Arm/Group | Dorsal Column Stimulation | Dorsal Root Ganglion Stimulation
Number analyzed (Participants) | 0 | 0

8. Other Pre Specified Outcome: Patients' Global Impression of Change (PGIC)
Description: Patients will be asked to rate their overall change in quality of health on a scale of 1 to 7 with 1 being no change in overall health and 7 being a great deal better in comparison to before implant. Another scale will on the same form ranging from 0-10 with 0 being much better, 5 being no change and 10 being much worse.
Time Frame: 6 Months
Population: Data were not collected
Arm/Group | Dorsal Column Stimulation | Dorsal Root Ganglion Stimulation
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Description: The definitions parallel those listed on clinicaltrials.gov
Arm/Group | Dorsal Column Stimulation | Dorsal Root Ganglion Stimulation
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-19): https://cdn.clinicaltrials.gov/large-docs/24/NCT03794024/Prot_SAP_000.pdf